CLINICAL TRIAL: NCT07212829
Title: Unravelling the Epigenetic Mechanisms of Exercise-induced Pain in Chronic Widespread Pain: DNA Methylation Regulation of the Brain-derived Neurotrophic Factor Expression and Its Modulation by Transcranial Direct Current Stimulation
Brief Title: The Added Value of Transcranial Direct Current Stimulation (tDCS) During Exercise for People With Chronic Widespread Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jo Nijs, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2025-255
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Widespread Pain; Fibromyalgia (FM)
Keywords: BDNF; pain; exercise; DNA methylation
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise + active tDCS + patients (Experimental): Patient participants will receive one bout of submaximal aerobic exercise, along with a single session of active tDCS simultaneously.
  Interventions: Device: Active tDCS; Behavioral: Aerobic exercise
- Exercise + sham tDCS + patients (Sham Comparator): Patient participants will receive one bout of submaximal aerobic exercise, along with a single session of sham tDCS simultaneously.
  Interventions: Behavioral: Aerobic exercise; Device: Sham tDCS
- Exercise + active tDCS + healthy controls (Active Comparator): healthy volunteer participants will receive one bout of submaximal aerobic exercise, along with a single session of active tDCS simultaneously.
  Interventions: Device: Active tDCS; Behavioral: Aerobic exercise
- Exercise + sham tDCS + healthy controls (Sham Comparator): healthy volunteer participants will receive one bout of submaximal aerobic exercise, along with a single session of sham tDCS simultaneously.
  Interventions: Behavioral: Aerobic exercise; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — tDCS is performed using a monophasic current device. Pairs of silicon sponge sur-face electrodes (35 cm2) are soaked in saline and positioned as follows: the anode is placed over the region of the dorsolateral prefrontal cortex (DLPFC) per the international 10/20 system at point F3 (left DLPFC), and the cathode is placed on the contralateral supraorbital area (FP2 site). For active tDCS, the current is ramped up for 30 seconds until the center electrode reaches a target intensity of 2 mA, then remains for 29 minutes before dropping for another 30s.
  Arms: Exercise + active tDCS + healthy controls; Exercise + active tDCS + patients
Behavioral: Aerobic exercise — Participants will perform a moderate aerobic exercise (AE, known as aerobic power index), using a cycle er-gometer. The exercise intensity is moderate and individually tailored based on each participant's estimated maximum heart rate (HRmax), calculated using the validated formula: HRmax = 211 - (0.64 × age).
Device: Sham tDCS — tDCS is performed using a monophasic current device. Pairs of silicon sponge sur-face electrodes (35 cm2) are soaked in saline and positioned as follows: the anode is placed over the region of the dorsolateral prefrontal cortex (DLPFC) per the international 10/20 system at point F3 (left DLPFC), and the cathode is placed on the contralateral supraorbital area (FP2 site).
  In the sham condition, current is ramped up to 2.0 mA for 30 seconds and then ramped down to 0 mA, with the total session duration matched to the active condition. This procedure was used to mimic the tingling sensa-tions typically experienced at the beginning of stimulation. Participants received identical instructions, session timing, and room setup across conditions.
  Arms: Exercise + sham tDCS + healthy controls; Exercise + sham tDCS + patients

SUMMARY:
Many people with chronic widespread pain (CWP) feel more pain and fatigue after exercise. This makes it hard to stay active. Unfortunately, the investigators do not fully understand why this happens and how to prevent it.

The primary goal of this study is to explore the underlying genetic and epigenetic mechanisms of BDNF gene in response to exercise, and investigate if transcranial direct current stimulation (tDCS) during exercise works to improve worsening symptoms response to exercise in people with CWP.

The investigators designed a randomized crossover study and will enroll 60 patients with CWP and 60 healthy controls. Participants will undergo 2 interventions in random order: 1) exercise + active tDCS, and 2) exercise + sham tDCS. Participants will visit the hospital twice with at least one week in between the visits.

DETAILED DESCRIPTION:
Many people with chronic widespread pain (CWP), such as those with fibromyalgia, experience increased pain in response to exercise, which discourages continued physical activity. Although abnormal gene expression via epigenetic mechanisms has been implicated in CWP, the underlying mechanisms by which exercise exacerbates symptoms remain unclear. DNA methylation is one way that environmental factors like exercise can alter gene expression, and brain-derived neurotrophic factor (BDNF) plays a central role in both neuroplasticity and pain processing. The investigators hypothesize that aberrant expression of the BDNF gene contributes to post-exercise symptom flares in CWP.

Transcranial direct current stimulation (tDCS) has been shown to modulate neuroplasticity and influence gene expression, making it a promising approach to normalize BDNF regulation during exercise.

In this randomized crossover trial, 60 CWP patients and 60 healthy controls will each undergo two sessions: (1) exercise with active tDCS and (2) exercise with sham tDCS. Each participant will visit the hospital twice, with at least one week between sessions. During each session, participants will receive one bout of submaximal aerobic exercise (20 min), along with a single session of active or sham tDCS (30 min) simultaneously. The order of interventions will be well-balanced and randomly allocated to each participant. We will measure pain intensity, serum BDNF protein levels, and BDNF gene methylation before and after each session. To capture longer-term effects, participants will also complete online symptom assessments at 8 hours, 24 hours, 48 hours, and 7 days post-exercise.

The primary objective of this study is to determine how active versus sham tDCS during exercise influences BDNF expression, DNA methylation patterns, and pain intensity in CWP patients.

The secondary objectives are to 1) compare these tDCS-induced changes between CWP patients and healthy controls; and 2) identify factors that influence tDCS/exercise-induced changes, including baseline BDNF levels, DNA methylation patterns, genetic polymorphisms and Lifestyle variables (e.g., physical activity).

By elucidating the epigenetic regulation of BDNF in exercise-induced pain and evaluating tDCS as a modulatory intervention, this study seeks to identify biomarkers of symptom exacerbation and develop non-pharmacological strategies that enable CWP patients to remain active without worsening their pain.

ELIGIBILITY:
Inclusion Criteria:

Patients

Participants in the patient group must meet all of the following criteria:

1. Diagnosis of chronic widespread pain (CWP) or fibromyalgia;
2. Age between 18 and 70 years old;
3. Body mass index (BMI) ≤ 35;
4. Widespread Pain Index (WPI) assessment: the WPI questionnaire (0-19 points) will be used to record the number and distribution of painful body sites. Participants will be classified as having CWP if pain is reported on both sides of the body, above and below the waist, and in the axial skeleton, with pain symptoms lasting ≥ 3 months;
5. Stable medication use for at least 1 month prior to study entry.

Healthy control group

Participants in the healthy control group must meet all of the following criteria:

1. Age between 18 and 70 years old;
2. Body mass index (BMI) ≤ 35;
3. No chronic conditions, such as chronic pain and diabetes.

Exclusion Criteria:

For both patients and healthy controls, participants will be excluded if they meet any of the following:

1. Current pregnancy or pregnancy within the past 12 months;
2. Contraindications for non-invasive brain stimulation (NIBS), in line with published safety guidelines;
3. History of neurological disorders, including epilepsy (personal or family history), traumatic brain injury, stroke, dementia, or Parkinson's disease;
4. Major medical conditions, including cancer, endocrine or metabolic disorders, urine, genital and cardiovascu-lar diseases (e.g., myocardial infarction, heart failure, arrhythmia, uncontrolled hypertension).
5. Substance abuse.
6. Presence of psychiatric disorders other than depression or anxiety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Participants rate their pain at baseline, and 30 minutes after the intervention.
  Pain intensity is measured using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no pain" and 10 indicates "the worst pain imaginable".
Blood BDNF levels | Blood samples are collected at baseline and 20 minutes after exercise-tDCS session.
  Venous blood samples are collected before and after each exercise-tDCS session. Samples are centrifuged, aliquoted, and stored at -80 °C until analysis. Blood levels of brain-derived neurotrophic factor (BDNF) are quantified using a commercially available enzyme-linked immunosorbent assay (ELISA), following the manufacturer's instructions.
BDNF DNA methylation | Blood samples are collected at baseline and 20 minutes after exercise-tDCS session.
  Genomic DNA is extracted from whole blood collected at baseline and after the intervention. DNA methylation of the BDNF gene is assessed using bisulfite conversion followed by quantitative analysis of methylation levels at CpG sites within promoter regions previously associated with pain regulation. Methylation levels are expressed as the percentage of methylated cytosines at each CpG site. Changes in DNA methylation are calculated as the difference between post-intervention and baseline values.

SECONDARY OUTCOMES:
Pain intensity | Participants rate their pain at immediately, 8 hours, 24 hours, 48 hours, and 7 days after the intervention.
  Pain intensity is measured using a 0-10 Numeric Rating Scale (NRS), where 0 indicates "no pain" and 10 indicates "the worst pain imaginable".
Fatigue | Participants rate their fatigue at baseline, and 24 hours, 48 hours, 7 days after the intervention.
  Brugmann Fatigue Scale (BFS). Fatigue is assessed with the BFS, an 8-item self-report questionnaire (4 mental and 4 physical items; each scored 0-3). Subscale scores range 0-12 (mental; physical), and the total score ranges 0-24; higher scores indicate greater fatigue/rest propensity.
Fibromyalgia symptom impact | Participants rate their FIQR at baseline, and 7 days after intervention.
  Revised Fibromyalgia Impact Questionnaire (FIQR). The FIQR evaluates the overall impact of fibromyalgia on functioning, symptoms, and quality of life. The total score ranges 0-100 (higher = greater disease burden), comprising function (0-30), overall impact (0-20), and symptoms (0-50) after standard weighting; each item is rated 0-10.
Central sensitization symptoms | Participants rate their CSI at baseline.
  The Central Sensitization Inventory (CSI) is administered to assess symptoms related to central sensitization, such as sensitivity to touch, light, or sound, sleep disturbances, and concentration difficulties. Scores range from 0 to 100, with higher scores reflecting greater symptom severity. Each item is rated 0-4.
Pain catastrophizing | Participants rate their PCS at baseline, and 30 minutes after the intervention.
  The Pain Catastrophizing Scale (PCS) is used to measure catastrophic thoughts and feelings related to pain, in-cluding rumination, magnification, and helplessness. Each item is rated 0-4. Total scores range from 0 to 52, with higher values indicating stronger pain catastrophizing tendencies.
Anxiety and depression | Participants rate their HAD at baseline.
  HADS consists of two subscales: HADS-A, designed to detect anxious states, and HADS-D, designed to detect de-pressive states. Each subscale consists of 7 items with a 4-point ordinal response format. Scores range from 0 to 21 in each subscale, with higher scores indicating higher levels of anxious or depressive state. Participants an-swer each item thinking of how they felt and/or behaved during the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- VUB, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Undecided